CLINICAL TRIAL: NCT05067699
Title: Serum Vitamin D Level Detection in Patients With Recurrent Pityriasis Versicolor
Brief Title: Vitamin D Level in Recurrent PV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Lecturer of Dermatology, faculty of Medicine, Cairo University., Kasr El Aini Hospital
Other Study IDs: VitD&PV
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Pityriasis Versicolor
MeSH Terms: conditions — Tinea Versicolor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients: recurrent pityriasis versicolor
  Interventions: Diagnostic Test: Human 25-Hydroxyvitamin D3 (HVD3) ELISA Kit (96 well)
- Controls: Healthy age and sex matched
  Interventions: Diagnostic Test: Human 25-Hydroxyvitamin D3 (HVD3) ELISA Kit (96 well)

INTERVENTIONS:
Diagnostic Test: Human 25-Hydroxyvitamin D3 (HVD3) ELISA Kit (96 well) — The serum will be tested by a double-antibody sandwich enzyme-linked immunosorbent assay (ELISA) to assay the level of Human 25Dihydroxy vitamin D（25-OH-D).

SUMMARY:
Serum Samples will be taken from patients with recurrent Pityriasis Versicolor for the evaluation of vitamin D level.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with recurrent pityriasis versicolor (active now) and not taking treatment for it.
* Patients of both genders.
* Age ≥18 years old.

Exclusion Criteria:

* - Patients with other cutaneous diseases.
* Patient's having dandruff (scaly scalp) even if not symptomatizing.
* Pregnant and lactating females, children, prisoners, cognitively impaired or mentally disabled subjects.
* Patients with autoimmune diseases.
* Patients with immunodeficiency diseases.
* Immunosuppressed patients e.g. HIV, diabetics, organ transplant, malignancy, patients taking immunosuppressive drugs e.g. chemotherapy, cortisone.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with recurrent Pityriasis Versicolor (more than 2 attacks per year) and of a disseminated nature
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum 25(OH) D3 level | 6months-1 year
  The serum of patients and controls will be tested by a double-antibody sandwich enzyme-linked immunosorbent assay (ELISA) to assay the level of Human 25Dihydroxy vitamin D（25-OH-D).

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Teaching Hospital, Cairo, Egypt